CLINICAL TRIAL: NCT01361048
Title: Neo-Penotran Forte Vaginal Suppository for Vaginal Trichomoniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Embil Pharmaceutical Co. Ltd (Industry)
Responsible Party: Principal Investigator, Jane Schwebke, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV-01
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Trichomonas Vaginitis
Keywords: trichomonas
MeSH Terms: conditions — Trichomonas Vaginitis; Trichomonas Infections | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- oral metronidazole (Active Comparator): control arm
  Interventions: Drug: oral metronidazole
- neo penotran forte (Experimental): neo penotran forte vaginal suppository twice a day for 7 days
  Interventions: Drug: neo penotran forte
- neo penotran forte once a day (Experimental): neo penotran forte vaginal suppository once a day for 7 days
  Interventions: Drug: neo penotran forte once a day

INTERVENTIONS:
Drug: oral metronidazole — 2 gm oral once
  Arms: oral metronidazole
Drug: neo penotran forte — neo penotran forte intravaginal twice a day for 7 days
  Arms: neo penotran forte
Drug: neo penotran forte once a day — neo penotran forte intravaginally once a day for 7 days
  Arms: neo penotran forte once a day

SUMMARY:
The investigators are trying a combination vaginal product of higher dose metronidazole combined with miconazole to see if it is effective in treating vaginal trichomonas.

ELIGIBILITY:
Inclusion Criteria:

* presence of trichomonas

Exclusion Criteria:

* pregnant or nursing
* known immunodeficiency
* allergy to study drugs
* concurrent yeast infection
* history of seizures or peripheral neuropathy
* unwillingness to abstain from alcohol during treatment period and for 48 hrs after concurrent lithium
* anticoagulation therapy, and abuse
* patient expected to have menses within 8 days of enrollment

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Personal Health Clinic UAB, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Metronidazole | Neo Penotran Forte | Neo Penotran Forte Once a Day
Started | 20 | 10 | 10
Completed | 20 | 10 | 9
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Neo Penotran Forte Twice a Day: neo penotran forte vaginal suppository twice a day for 7 days
- Total: Total of all reporting groups
Arm/Group | Oral Metronidazole | Neo Penotran Forte Twice a Day | Neo Penotran Forte Once a Day | Total
Number analyzed (Participants) | 20 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (11.8) | 31.5 (9.8) | 28.3 (6.7) | 30.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 10 | 40
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Cured of Vaginal Trichmonas
Description: percentage of participants achieving microbiological cure of trichomonas
Time Frame: day 12-15
Measure: Number; unit: percentage of participants
Groups:
- Oral Metronidazole 2 gm Stat Dose: control arm
Arm/Group | Oral Metronidazole 2 gm Stat Dose | Neo Penotran Forte | Neo Penotran Forte Once a Day
Number analyzed (Participants) | 20 | 10 | 9
percentage of participants | 90 | 90 | 88

2. Secondary Outcome: Tolerability of the Study Product as Measured by Participant Self-report
Description: Number of participants with any side effects
Time Frame: day 12-15 day 30-35
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Metronidazole | Neo Penotran Forte | Neo Penotran Forte Once a Day
Number analyzed (Participants) | 20 | 10 | 9
Participants | 2 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Oral Metronidazole | Neo Penotran Forte | Neo Penotran Forte Once a Day
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/20 | 1/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Metronidazole (N=20) | Neo Penotran Forte (N=10) | Neo Penotran Forte Once a Day (N=10)
suicicdal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Metronidazole (N=20) | Neo Penotran Forte (N=10) | Neo Penotran Forte Once a Day (N=10)
vaginal itch (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No